CLINICAL TRIAL: NCT02605200
Title: Identification and Treatment of Diabetes In Solid Organ Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jee-Young Nina Ham, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00081257
Record Dates: First submitted 2015-10-06; First posted 2015-11-16 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Complications of Transplanted Organs and Tissue
Keywords: Diabetes; Endocrinology; Pediatrics
MeSH Terms: conditions — Diabetes Mellitus | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): Participants will complete tests of glucose tolerance and psychosocial assessments, and will undergo medical history screening. Those children identified with diabetes and/or abnormal glucose tolerance will receive both diabetes self-management education and psychosocial support from a pediatric Certified Diabetes Educator (CDE) and a psychologist, respectively.
  Interventions: Behavioral: Psychologist Support; Behavioral: Pediatric Certified Diabetes Educators (CDEs) Support

INTERVENTIONS:
Behavioral: Psychologist Support — Participants will complete several psychological questionnaires that are intended to cover a broad spectrum of physical, mental, and emotional aspects of the health of participants; the Behavior Assessment System for Children (BASC) ,the Children Depression Inventory (CDI 2), the Pediatric Quality of Life Inventory Transplant Module (PedsQL), and the Wechsler Abbreviated Scale of Intelligence II (WASI-II). Data gathered from this testing will be used to guide the provision of psychological care to address psychosocial challenges inherent to the care of children with transplant related diabetes.
Behavioral: Pediatric Certified Diabetes Educators (CDEs) Support — Pediatric Certified Diabetes Educators (CDEs) are specially trained to teach diabetes self-management to children and their families. Participants who are diagnosed with diabetes will receive individualized support from a CDE in conjunction with their routine transplant care.

SUMMARY:
The purpose of this study is to determine the influence of post-transplant diabetes on medical and psychosocial outcomes in individuals who receive solid-organ transplant prior to 18 years of age and their families.

DETAILED DESCRIPTION:
This study seeks to understand how organ transplant patients are affected by the development of diabetes, and to test whether early diagnosis of diabetes and comprehensive professional support will:

1. facilitate the adjustment of children and their families to the rigors of diabetes care
2. improve adherence to medication regimens
3. reduce acute complications of diabetes and organ rejection.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Children's Healthcare of Atlanta who have received a kidney, liver, or heart transplant

Exclusion Criteria:

* Received a transplant after 18 years of age
* Cognitively unable to participant as determined by the study team psychologist
* Not receiving a solid organ transplant for kidney, liver, or heart
* Declines participation invitation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Change in the Pediatric Quality of Life Inventory Transplant Module (PedsQL) | Baseline, interval, and end of participation (Up to 18 years of age)
  The Pediatric Quality of Life Inventory Transplant Module (PedsQL) is a 15 minute survey intended to measure emotional and physical function in children and determine state of wellbeing.

SECONDARY OUTCOMES:
Transplant Rejection Rate Post Diabetes Diagnosis | Up to three years
  Participants will be followed at Children's Healthcare of Atlanta, and monitored for rates of transplant rejection after being diagnosed with diabetes.
Rate of Vascular Disease Post Diabetes Diagnosis | Up to three years
  Participants will be followed at Children's Healthcare of Atlanta, and monitored for rates of vascular disease after being diagnosed with diabetes.
Mortality Rate Post Diabetes Diagnosis | Up to three years
  Participants will be followed at Children's Healthcare of Atlanta, and monitored for rates of mortality after being diagnosed with diabetes.
Change in the Wechsler Abbreviated Scale of Intelligence II (WASI-II) Score | Baseline, interval, and end of participation (Up to 18 years)
  The Wechsler Abbreviated Scale of Intelligence II (WASI-II) is intended to determine cognitive ability for use in educational, as well as clinical and research settings. The WASI-II is ideal for any subject over the age of six, and takes approximately one hour to complete.
Change in the Children Depression Inventory (CDI 2) Score | Baseline, interval, and end of participation (Up to 18 years)
  The Children Depression Inventory (CDI 2) is a short ten minute self-reported survey intended to aid in the assessment of signs of depression in children ages seven through 17. This test helps determine negative mood, poor self-esteem, a loss of interest in activities, interpersonal problems, and feelings of ineffectiveness, the common traits of depression.
Change in the Behavior Assessment System for Children (BASC) Score | Baseline, interval, and end of participation (Up to 18 years)
  The Behavior Assessment System for Children (BASC) takes approximately 15 minutes to complete and is intended to determine emotional and behavioral change in children, as well as to indicate risks to their health and development

CONTACTS AND LOCATIONS:
Overall Officials: Nina Ham, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia